CLINICAL TRIAL: NCT03157193
Title: Effect of Hyaluronic Acid on Peri-implant Pathology: A Double-blind, Randomized, Controlled Clinical Trial.
Brief Title: Effect of Hyaluronic Acid on Perimplantitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Ricerfarma S.r.l (Other)
Responsible Party: Principal Investigator, Francisco Mesa, Associate Professor in Periodontology, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OTRI-3300
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis; Dental Implants; Hyaluronic Acid; Clinical Trial
MeSH Terms: conditions — Peri-Implantitis | interventions — Hyaluronic Acid; hydroxypropyl guar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Group (Experimental): Hyaluronic acid gel 0.2% at baseline and later home applications by the patients during 45 days.
  Interventions: Drug: Hyaluronic Acid
- Control 1 Group (Sham Comparator): Hydroxypropyl guar based gel, without any biological effect.
  Interventions: Drug: Hydroxypropyl Guar
- Control 2 Group (No Intervention): No gel application, only standard perimplantitis treatment.

INTERVENTIONS:
Drug: Hyaluronic Acid — Hyaluronic acid gel application as coadjuvant in the treatment of perimplantitis.
  Other Names: HA
  Arms: Test Group
Drug: Hydroxypropyl Guar — Hydroxypropyl Guar gel application as sham comparator
  Other Names: Control 1
  Arms: Control 1 Group

SUMMARY:
The effect of the hyaluronic acid treatment on peri-implantitis has not been tested. The aim was to analyze the effect of a hyaluronic acid-containing gel on the clinical variables and the expression of biochemical inflammatory markers in the crevicular fluid of implants receiving perimplantitis treatment.

DETAILED DESCRIPTION:
The aim was to analyze the effect of a hyaluronic acid-containing gel on the clinical variables and the expression of biochemical inflammatory markers in the crevicular fluid of implants receiving perimplantitis treatment.

A randomized, controlled, double-blind clinical trial was designed on 100 perimplantitis affected implants placed in 61 subjects. Inclusion criteria were implants with at least 1 year of functional loading and with diagnosis of perimplantitis following the criteria from the Association of Dental Implantology. All implant received perimplantitis treatment. Each patient was randomly assigned to receive a gel containing 0.8% HA (Test group), a gel without HA (Placebo group) or no gel treatment (Control group). After a first gel application at baseline, test and placebo patients performed gel applications at home 3 times/day for 45 days. Clinical variables of each implant were recorded at baseline, 45 and 90 days (probing depth, attachment loss, bleeding). Intraoral radiographs of each implants were performed to measure marginal bone level. Peri-implant crevicular fluid was collected from each implant at baseline and after 45 days of treatment, to assess IL-1β and TNFα levels by ELISA technique. Clustering analysis, considering multiple implants within each patient, was performed.

ELIGIBILITY:
Inclusion Criteria:

* Implants with at least one year of functional load.
* Implants diagnosed with peri-implantitis according to the criteria of the Association of Dental Implantology.

Exclusion Criteria:

* Previous peri-implantitis treatment.
* Pregnancy or breast-feeding.
* Neoplastic disease.
* Antibiotic treatment during the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Peri-implant probing depth | Baseline, change at 45 days and at 90 days.
  Probing depth (mm) assessed by periodontal probe.
Peri-implant attachment level | Baseline, change at 45 days and at 90 days.
  Probing attachment level (mm) calculated using probing depth and exposed implant threads.
Peri-implant bleeding | Baseline, change at 45 days and at 90 days.
  Bleeding on probing expressed as % of bleeding implants in each group.
Marginal Bone level | Baseline, change at 45 days and at 90 days.
  Alveolar bone level assesed in periapical digital radiographs by image processing software (ImageJ).
Peri-implant crevicular fluid cytokines. | Baseline and change at 45 days.
  Inflammatory cytokines (IL1B and TNFa) measured in Peri-implant crevicular fluid by ELISA.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Fernandez E, Magan-Fernandez A, O'Valle F, Bravo M, Mesa F. Hyaluronic acid reduces inflammation and crevicular fluid IL-1beta concentrations in peri-implantitis: a randomized controlled clinical trial. J Periodontal Implant Sci. 2021 Feb;51(1):63-74. doi: 10.5051/jpis.1903660183. PMID 33634616